CLINICAL TRIAL: NCT00322179
Title: Microarray Analysis of IFN-Induced Gene Expression in Obese and Non-Obese Patients With Chronic Hepatitis C
Status: Completed | Type: Observational
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Principal Investigator, Ramsey Cheung, Principal Investigator, Palo Alto Veterans Institute for Research
Other Study IDs: CHR0036ARG; PEG215
Record Dates: First submitted 2006-05-04; First posted 2006-05-05 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Hepatitis C; Obesity
Keywords: Microarray Analysis; Obesity; Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other

GROUPS / COHORTS (2):
- Obese
- Non-Obese

SUMMARY:
The response rate to interferon-based anti-viral therapy for chronic hepatitis C is lower in patients who are obese. However, it is not clear whether this is related to suboptimal dosing of the medication or alterated response in obese patients. Alterated immune response had been reported in obese patients. The goal of current study is to determine the immune response to interferon in obese compared to non-obese chronic hepatitis C in an tissue culture system.

DETAILED DESCRIPTION:
To examine our hypothesis, we will incubate PBMC samples from obese and nonobese patients with IFN, followed by microarray analysis to compare the IFN response patterns in both groups of patients and to identify genes differentially regulated between these two groups. Identification of such genes will provide important insight to the mechanism of the antiviral effect of HCV. The identified genes will have the potential of serving as targets for pharmaceutical intervention aiming at enhancing the efficacy of IFN therapy for obese patients.

This is an open-label study. Ten obese and 10 nonobese patients with chronic hepatitis C will be recruited. For the purpose of this study, obese is defined as body weight >85 kg and BMI >30, and nonobese as body weight <75 kg and BMI<25.

ELIGIBILITY:
Inclusion Criteria:

* obese (weight > 85kg and BMI>30) or non-obese patients (<75kg and BMI <25) with chronic Hepatitis C
* Chronic Hepatitis C infection with documented HCV RNA
* Body habitat either as obese or non-obese as defined above
* Currently not under IFN therapy
* Non-African American

Exclusion Criteria:

* Body habitat neither obese or non-obese as defined for the purpose of this study
* Unable to give consent
* On immunomodulatory agents such as prednisone
* Active infection other than Hepatitis C
* Co-infection with HBV or HIV
* Active or excessive alcohol use
* Other cause of chronic Hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * obese (weight > 85kg and BMI>30) or non-obese patients (<75kg and BMI <25) with chronic Hepatitis C
  * Chronic Hepatitis C infection with documented HCV RNA
  * Body habitat either as obese or non-obese as defined above
  * Currently not under IFN therapy
  * Non-African American
Enrollment: 22 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramsey Cheung, MD, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] Bressler BL, Guindi M, Tomlinson G, Heathcote J. High body mass index is an independent risk factor for nonresponse to antiviral treatment in chronic hepatitis C. Hepatology. 2003 Sep;38(3):639-44. doi: 10.1053/jhep.2003.50350. PMID 12939590
- [Background] Camps J, Crisostomo S, Garcia-Granero M, Riezu-Boj JI, Civeira MP, Prieto J. Prediction of the response of chronic hepatitis C to interferon alfa: a statistical analysis of pretreatment variables. Gut. 1993 Dec;34(12):1714-7. doi: 10.1136/gut.34.12.1714. PMID 7904252
- [Background] Farooqi IS, Matarese G, Lord GM, Keogh JM, Lawrence E, Agwu C, Sanna V, Jebb SA, Perna F, Fontana S, Lechler RI, DePaoli AM, O'Rahilly S. Beneficial effects of leptin on obesity, T cell hyporesponsiveness, and neuroendocrine/metabolic dysfunction of human congenital leptin deficiency. J Clin Invest. 2002 Oct;110(8):1093-103. doi: 10.1172/JCI15693. PMID 12393845
- [Background] Fried MW, Shiffman ML, Reddy KR, Smith C, Marinos G, Goncales FL Jr, Haussinger D, Diago M, Carosi G, Dhumeaux D, Craxi A, Lin A, Hoffman J, Yu J. Peginterferon alfa-2a plus ribavirin for chronic hepatitis C virus infection. N Engl J Med. 2002 Sep 26;347(13):975-82. doi: 10.1056/NEJMoa020047. PMID 12324553
- [Background] Ji X, Cheung R, Cooper S, Li Q, Greenberg HB, He XS. Interferon alfa regulated gene expression in patients initiating interferon treatment for chronic hepatitis C. Hepatology. 2003 Mar;37(3):610-21. doi: 10.1053/jhep.2003.50105. PMID 12601359